CLINICAL TRIAL: NCT01429649
Title: A Prospective Study of Ablation of Pulmonary Focal Pure Ground Glass Opacity
Brief Title: Study of Ablation for the Pulmonary Focal Pure Ground Glass Opacity (pGGO)
Acronym: pGGO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chen Weisheng, The vice chief of the Thoracic Division, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kj2011001
Record Dates: First submitted 2011-09-03; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Pulmonary Lesions
Keywords: pure pulmonary ground glass opacity
MeSH Terms: interventions — Cryotherapy; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ablation (Experimental): Cryoablation or Radiofrequency ablation for the pGGO
  Interventions: Procedure: cryotherapy or radiofrequency ablation
- Follow up CT scann (No Intervention): The patients will receive follow up with CT scan every 6-9 months.

INTERVENTIONS:
Procedure: cryotherapy or radiofrequency ablation — Cryoablation or Radiofrequency ablation is performed under CT image guidance.
  Arms: ablation

SUMMARY:
With the advent of CT screening for lung cancer, there is an increase in the detection of pulmonary lesions with focal pure ground-glass opacity (pGGO). The pure Ground-glass opacities can be caused by normal expiration, partial filling of air spaces, partial collapse of alveoli, interstitial thickening, inflammation, oedema, fibrosis, and lepidic proliferation of neoplasm. Precise details of the natural history of focal pure GGO are still largely unclear. A number of differential diagnoses are possible, including inflammatory disease, focal scar, atypical adenomatous hyperplasia (AAH), and adenocarcinoma in situ. Some of pGGOs remained stable over a considerable time. A long doubling time for pGGOs is already known. Therefore, the strategy of treatment for focal pure GGO lesions is still undecided. The major issue is whether or not the doctors should treat these patients at all or wait until the first sign of a solid lesion developes which may take many years.

The purpose of this study is to determine if the ablation therapy is safe and effective for the pulmonary pGGO.

ELIGIBILITY:
Inclusion Criteria:

* The lesion(s) treated with ablation must be =< 2.0 cm in greatest dimension
* All patients are required to have been evaluated in a multi-disciplinary tumor conference to ensure that the lesion is suitable for Image-guided percutaneous ablation
* Platelet count ≥ 100 x 109/L
* International normalized ratio (INR) < 1.5
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* A signed study specific consent form is required

Exclusion Criteria:

* Direct evidence of regional or distant metastases,or synchronous primary or prior malignancy in the past 5 years
* Unable to lie flat or has respiratory distress at rest
* Uncontrolled coagulopathy or bleeding disorders
* Evidence of active systemic, pulmonary, or pericardial infection
* Women who are pregnant or breastfeeding
* Patients with poor pulmonary function

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The changing of the lesion | 3 years
  To determine the efficacy rate of CT image guided ablation for pulmonary focal pGGO.
  To determine the feasibility and safety of CT image guided ablation in patients with pulmonary pGGO.

SECONDARY OUTCOMES:
The side effect of the therapy. | 3 years
  Intra and post-operative complications rates. Quality-of-life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Weisheng Chen, MD, Principal Investigator — Dongfang Hospital Beijing University of Chinese Medicine
Locations (1):
- Dongfang Hospital, Fuzhou, Fujian, China